CLINICAL TRIAL: NCT07000149
Title: A Phase Ib/III Randomized, Multicenter, Global Study of Volrustomig Plus Casdatifan or Volrustomig Monotherapy Versus Nivolumab Plus Ipilimumab as First-line Treatment for Participants With Advanced Clear Cell Renal Cell Carcinoma (ccRCC)
Brief Title: A Study to Investigate the Efficacy and Safety of Volrustomig ± Casdatifan vs Nivolumab + Ipilimumab as 1L Treatment for Advanced ccRCC
Acronym: eVOLVE-RCC02
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D798NC00001; 2024-519865-23-00 (Other: EU CT Number)
Record Dates: First submitted 2025-05-23; First posted 2025-06-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma
Keywords: Programmed cell death-ligand-1; Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4); First-line treatment (1L); Immunotherapy; Kidney cancer; Clear cell renal carcinoma; Immuno-oncology bispecific (IO-bispecific); Volrustomig; Casdatifan; Hypoxia-inducible factor-2α (HIF-2α)
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12; Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1A (Volrustomig Dose 1 + Casdatifan) (Experimental): Participants will receive dose 1 of volrustomig in combination with casdatifan.
  Interventions: Drug: Volrustomig; Drug: Casdatifan
- Arm 1B (Volrustomig Dose 2 + Casdatifan) (Experimental): Participants will receive dose 2 of volrustomig in combination with casdatifan.
  Interventions: Drug: Volrustomig; Drug: Casdatifan
- Arm 3A (Volrustomig Dose X + Casdatifan) (Experimental): Participants will receive Volrustomig at the dose to be determined in the Phase Ib part of the study, in combination with casdatifan.
  Interventions: Drug: Volrustomig; Drug: Casdatifan
- Arm 3B (Volrustomig Dose 1) (Experimental): Participants will receive dose 1 of volrustomig.
  Interventions: Drug: Volrustomig
- Arm 3C (Nivolumab + Ipilimumab) (Active Comparator): Participants will receive nivolumab plus ipilimumab as standard of care treatment.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Volrustomig — Volrustomig will be administered as an intravenous (IV) infusion.
  Other Names: MEDI5752
  Arms: Arm 1A (Volrustomig Dose 1 + Casdatifan); Arm 1B (Volrustomig Dose 2 + Casdatifan); Arm 3A (Volrustomig Dose X + Casdatifan); Arm 3B (Volrustomig Dose 1)
Drug: Casdatifan — Casdatifan will be administered orally.
  Other Names: AB521
  Arms: Arm 1A (Volrustomig Dose 1 + Casdatifan); Arm 1B (Volrustomig Dose 2 + Casdatifan); Arm 3A (Volrustomig Dose X + Casdatifan)
Drug: Nivolumab — Nivolumab will be administered as an IV infusion.
  Other Names: Opdivo
  Arms: Arm 3C (Nivolumab + Ipilimumab)
Drug: Ipilimumab — Ipilimumab will be administered as an IV infusion.
  Other Names: Yervoy
  Arms: Arm 3C (Nivolumab + Ipilimumab)

SUMMARY:
This is a Phase Ib/III, randomized, multicenter, global study evaluating the efficacy and safety of volrustomig in combination with casdatifan for the first-line (1L) treatment of participants with advanced clear cell renal cell carcinoma (ccRCC).

DETAILED DESCRIPTION:
The primary purpose of this study is to determine the recommended Phase III dose (RP3D) of volrustomig and measure the efficacy and safety of volrustomig in combination with casdatifan compared with nivolumab plus ipilimumab in participants with advanced ccRCC (as 1L treatment).

The study comprises of 2 parts -

In Phase 1b part of the study, participants will be randomized in a 1:1 ratio to receive either dose 1 or dose 2 of volrustomig in combination with casdatifan.

In Phase III part of the study, participants will be randomized in 1:1:1 to receive either Volrustomig (at the dose to be determined in the Phase Ib) in combination with casdatifan, volrustomig monotherapy or standard of care (nivolumab plus ipilimumab).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed RCC with clear cell component.
* Advanced/metastatic RCC or recurrent disease that has not previously been treated with systemic therapy in the 1L setting.
* Karnofsky Performance Status ≥ 70%.
* Provision of acceptable tumor sample.
* At least one lesion that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and is suitable for accurate repeated measurements.

Exclusion Criteria:

* History of leptomeningeal disease or spinal cord compression.
* Symptomatic brain metastases.
* Medical history of severe chronic obstructive pulmonary disease.
* Active or prior documented autoimmune or inflammatory disorders.
* Prior systemic therapy for advanced/metastatic RCC. Note - Other inclusion and exclusion criteria may apply as stated in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2030-02-21 (Estimated); Study Completion 2032-07-29 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Approximately 39 months
  Number of participants who received at least one dose of study treatment will be assessed.
Phase III: Progression-free Survival (PFS) | Approximately 38 months
  The PFS is defined as the time from randomization until radiological progression or death due to any cause (in the absence of progression).
Phase III: Overall Survival (OS) | Approximately 67 months
  The OS is defined as the time from randomization until the date of death due to any cause.

SECONDARY OUTCOMES:
Phase Ib: Objective Response rate (ORR) | Approximately 39 months
  The ORR is defined as the proportion of participants who have a confirmed complete response (CR) or confirmed partial response (PR).
Phase Ib: Duration of Response (DoR) | Approximately 39 months
  The DoR is defined as the time from the date of first documented confirmed response until date of documented progression or death due to any cause.
Phase Ib: Progression-free Survival (PFS) | Approximately 39 months
  The PFS is defined as the time from randomization until radiological progression or death due to any cause (in the absence of progression).
Phase Ib: Disease Control Rate (DCR) | Approximately 39 months
  The DCR is defined as the percentage of participants who have a confirmed CR or PR or who have stable disease (SD) after randomization.
Phase Ib: Volrustomig concentration in serum | Up to 27 months
  To assess the serum concentration of volrustomig when administered concomitantly with casdatifan.
Phase Ib: Casdatifan concentration in plasma | Up to 27 months
  To assess the plasma concentration of casdatifan when administered concomitantly with volrustomig.
Phase Ib: Time to Response (TTR) | Approximately 39 months
  The TTR is defined as the time from randomization until the first documentation of a subsequently confirmed objective response.
Phase III: Overall Survival | Approximately 67 months
  The OS is defined as the time from randomization until the date of death due to any cause.
Phase III: Number of participants with AEs and SAEs | Approximately 67 months
  Number of participants who received at least one dose of study treatment will be assessed.
Phase III: Time to second progression or death (PFS2) | Approximately 67 months
  The PFS2 is defined as the time from randomization to the earliest progression event after the start of the first subsequent therapy, or death from any cause, whichever occurs first.
Phase III: Objective Response rate (ORR) | Approximately 67 months
  The ORR is defined as the proportion of participants who have a confirmed CR or confirmed PR.
Phase III: Duration of Response (DoR) | Approximately 67 months
  The DoR is defined as the time from the date of first documented confirmed response until date of documented progression or death due to any cause.
Phase III: Progression-free Survival | Approximately 67 months
  The PFS is defined as the time from randomization until radiological progression or death due to any cause (in the absence of progression).

CONTACTS AND LOCATIONS:
Locations (25):
- United States (7):
  - Research Site, La Jolla, California
  - Research Site, Aurora, Colorado
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Lubbock, Texas
- Australia (4):
  - Research Site, East Melbourne
  - Research Site, Elizabeth Vale
  - Research Site, North Adelaide
  - Research Site, Syndey
- China (6):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Xiamen
- Georgia (2):
  - Research Site, Batumi
  - Research Site, Tbilisi
- South Korea (3):
  - Research Site, Busan
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/